CLINICAL TRIAL: NCT01069900
Title: A Randomized, Double-blind, Multicenter Trial to Evaluate the Safety and Efficacy of Sequential (Intravenous, Oral) Moxifloxacin Versus Comparator in Pediatric Subjects With Complicated Intra-abdominal Infection
Brief Title: Moxifloxacin in Pediatric Subjects With Complicated Intra-abdominal Infection
Acronym: MOXIPEDIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11643; 1962 (Avelox pediatrics) (Other: Company internal); 2009-015578-37 (EudraCT Number)
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Intraabdominal Infections
Keywords: Intra-abdominal infection; Pediatric infection
MeSH Terms: conditions — Intraabdominal Infections | interventions — Moxifloxacin; Ertapenem; Amoxicillin-Potassium Clavulanate Combination; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Avelox, BAY12-8039) (Experimental): Subjects randomized to the moxifloxacin arm of this study received intravenous moxifloxacin plus ertapenem placebo (0.9 % sodium chloride [NaCl solution]) for a minimum of 3 days and, if switched to oral treatment, PO moxifloxacin plus PO amoxicillin/clavulanate placebo. Total treatment duration is 5-14 days.
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039); Drug: Ertapenem placebo; Drug: Amoxicillin/Clavulanate placebo
- Comparator Ertapenem (Active Comparator): Subjects randomized to the comparator arm of this study received intravenous ertapenem plus moxifloxacin placebo (0.9 % NaCl solution) for a minimum of 3 days and, if switched to oral treatment, amoxicillin/clavulanate as an oral suspension plus PO moxifloxacin placebo. Total treatment duration is 5-14 days.
  Interventions: Drug: Ertapenem; Drug: Amoxicillin/Clavulanate; Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — For subjects 12 to less than (<) 18 years of age and weighing at least 45 kilograms (kg), the dose of moxifloxacin will be 400 milligrams (mg), once daily (OD). Subjects 12 to < 18 years of age and weighing less than 45 kg, the dose of moxifloxacin will be 4 mg/kg twice daily (BID), every 12 hours (q12h), not exceeding 400 mg/day. Subjects 6 to < 12 years of age the dose of moxifloxacin will be 4mg/kg, q12h, not exceeding 400 mg/day. Subjects 2 to less than 6 years of age the dose of moxifloxacin will be 5mg/kg, q12h, not exceeding 400 mg/day. Subjects 3 months to less than 2 years of age the dose of moxifloxacin will be 6mg/kg q12h IV, not exceeding 400 mg/day. Subjects who were switched from IV to PO therapy, 400 mg or 50 mg moxifloxacin tablets were provided.
  Arms: Moxifloxacin (Avelox, BAY12-8039)
Drug: Ertapenem — For subjects 13 to <18 years of age, the dosage of ertapenem was 1 gram (g) OD. For subjects 3 months to < 13 years of age, the dosage was 15 mg/kg q12h not to exceed 1 g/day.
  Arms: Comparator Ertapenem
Drug: Amoxicillin/Clavulanate — Subjects 2 years to < 18 years of age who were switched from IV to PO therapy receive amoxicillin/clavulanate suspension. The dosage of clavulanate was 3.2 mg/kg q12h. (maximum dose of clavulanate was 125 mg q12h). The dosage of amoxicillin was 22.5 mg q12h (a maximum dose of 875 mg amoxicillin q12h must not be exceeded).
  Arms: Comparator Ertapenem
Drug: Moxifloxacin placebo — Sterile 0.9% sodium chloride solution intended for IV use was used as the placebo for IV moxifloxacin. Tablets containing inactive ingredients were used as the placebo for PO moxifloxacin 400 mg and 50 mg tablets.
  Arms: Comparator Ertapenem
Drug: Ertapenem placebo — Sterile 0.9% sodium chloride solution intended for IV use was used as the placebo for IV ertapenem.
  Arms: Moxifloxacin (Avelox, BAY12-8039)
Drug: Amoxicillin/Clavulanate placebo — Suspension containing inactive ingredients was used as the placebo for PO amoxicillin/clavulanate suspension.
  Arms: Moxifloxacin (Avelox, BAY12-8039)

SUMMARY:
The primary focus of the study is the evaluation of the safety of treatment with moxifloxacin in a pediatric population 3 months to <18 years old. Approximately 450 pediatric subjects with a complicated intra-abdominal infection will be enrolled in the study and treated with either moxifloxacin intravenously and orally if switched to oral therapy or ertapenem (intravenously) and, if switched to oral therapy, amoxicillin/clavulanate.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized males or females 3 months to 17 years of age
* Able to obtain parental or legal guardian written informed consent and assent from subjects as applicable by local laws and regulations
* Expected duration of treatment with antibiotics is a minimum of 3 days administered IV, for a total of 5 to 14 days administered IV or IV followed by PO
* If the subject is a female of child-bearing potential she must have a negative pregnancy test at the screening visit or be capable of practicing an adequate method of contraception, and agree to continue the same method for 1 month following the TOC visit. Lactating subjects are not to be included.
* Subjects may be enrolled upon a surgically (laparotomy, laparoscopy, or percutaneous drainage) confirmed cIAI revealing at least one of the following:

  * Gross peritoneal inflammation with purulent exudate within the abdominal cavity
  * Intra-abdominal abscess
  * Macroscopic intestinal perforation with diffuse peritonitis OR
* Subjects may be enrolled on the basis of a suspected cIAI, which must be supported with radiological evidence (ultrasound, abdominal plain films, computed tomography [CT], magnetic resonance imaging [MRI]) of gastrointestinal perforation or localized collections of potentially infected material and at least one of the following:

  * Symptoms referable to the abdominal cavity (eg, anorexia, nausea, vomiting or pain)
  * Tenderness (with or without rebound), involuntary guarding, absent or diminished bowel sounds, or abdominal wall rigidity
  * Fever
  * Leukocytosis
* The subject must be scheduled for a surgical procedure (laparotomy or laparoscopy) or percutaneous drainage.

Exclusion Criteria:

* Presumed spontaneous bacterial peritonitis
* All pancreatic processes including pancreatic sepsis, peripancreatic sepsis, or an cIAI secondary to pancreatitis
* Early acute or suppurative (nonperforated) appendicitis unless there is evidence of an abscess or peritoneal fluid containing pus and micro-organisms suggestive of regional contamination
* Infections originating from the female genital tract
* Known severe immunosuppression. Subjects with known mild immunosuppression (eg, Type I or II diabetes mellitus, trauma, or absolute neutrophil count [ANC] between 1000 and 1500 cells/mm3) may be enrolled.
* Congenital or documented acquired QT prolongation
* Receiving concomitant treatment with QT prolonging drugs
* History of tendon disease/disorder related to quinolone treatment
* Pathogenic organisms suspected or identified (eg, Pseudomonas) which are resistant to any of the study drugs
* Abnormal musculoskeletal findings at baseline assessment; or chronic musculoskeletal disease (eg, juvenile rheumatoid arthritis); or chronic illness with high risk for chronic or recurrent arthritis or tendinitis (eg, cystic fibrosis, chronic inflammatory bowel disease)
* History of myasthenia gravis

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 458 (Actual)
Dates: Start 2010-07-21 (Actual); Primary Completion 2015-01-21 (Actual); Study Completion 2015-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (38):
- United States (2):
  - San Diego, California
  - Springfield, Massachusetts
- Hospital de Agudos "Dr. Carlos Bocalandro", Tres de Febrero, Buenos Aires, Argentina
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
- Canada (3):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Montreal, Quebec
- Santiago, Chile
- Czechia (2):
  - Olomouc
  - Prague
- Germany (3):
  - Stuttgart, Baden-Wurttemberg
  - Regensburg, Bavaria
  - Wuppertal, North Rhine-Westphalia
- Athens, Greece
- Hungary (2):
  - Budapest
  - Győr
- Latvia (3):
  - Daugavpils
  - Rēzekne
  - Riga
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (3):
  - Guadalajara, Jalisco
  - México, D.F., Mexico City
  - Ecatepec de Morelos, State of Mexico
- Peru (2):
  - Cusco
  - Lima
- Romania (2):
  - Iași
  - Timișoara
- Russia (2):
  - Smolensk
  - Vladikavkaz
- Ukraine (4):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Lviv
  - Simferopol

REFERENCES:
- [Result] Wirth S, Emil SGS, Engelis A, Digtyar V, Criollo M, DiCasoli C, Stass H, Willmann S, Nkulikiyinka R, Grossmann U; MOXIPEDIA Study Group. Moxifloxacin in Pediatric Patients With Complicated Intra-abdominal Infections: Results of the MOXIPEDIA Randomized Controlled Study. Pediatr Infect Dis J. 2018 Aug;37(8):e207-e213. doi: 10.1097/INF.0000000000001910. PMID 29356761
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multicenter between 21 July 2010 (first subject first visit) to 21 January 2015 (last subject last visit).
Pre-assignment Details: Overall 478 subjects were enrolled, 20 subjects had screening failures hence, 458 subjects were randomized to receive treatment.
Groups:
- Moxifloxacin (Avelox, BAY12-8039): Subjects randomized to the moxifloxacin arm of this study received intravenous moxifloxacin plus ertapenem placebo (0.9 % sodium chloride [NaCl solution]) for a minimum of 3 days and, if switched to oral treatment, PO moxifloxacin plus PO amoxicillin/clavulanate placebo. Total treatment duration is 5- 14 days.
Period: Overall Study
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Started | 305 | 153
Treated | 301 | 150
Completed | 287 | 149
Not Completed | 18 | 4
Not completed — Technical problems | 0 | 1
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Insufficient Therapeutic effect | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem | Total
Number analyzed (Participants) | 305 | 153 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.05 (3.66) | 12.046 (3.495) | 12.049 (3.602)
Age, Customized [Number; unit: Subjects]
  12 - < 18 years | 190 | 94 | 284
  6 - < 12 years | 100 | 52 | 152
  2 - < 6 years | 14 | 7 | 21
  3 months - < 2 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 53 | 177
  Male | 181 | 100 | 281

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: All AEs and SAE were recorded from treatment start to test of cure visit; musculoskeletal AEs were recorded up to 1 year post-end of treatment (EOT) visit; subjects with musculoskeletal AEs 1 year after EOT were followed up to 5 years or until resolution.
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number; unit: Subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Subjects
  Any AE | 175 | 82
  Any SAE | 20 | 6

2. Primary Outcome: Number of Subjects With Clinical Cardiac Adverse Events
Time Frame: Clinical cardiac event related to QT interval were recorded from treatment start until day 3 of treatment. All other clinical cardiac events were recorded from treatment start to test of cure visit, up to day 56.
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number; unit: Subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Subjects
  Any AE | 38 | 7
  Any SAE | 0 | 0

3. Primary Outcome: Number of Subjects With Musculoskeletal Adverse Events
Time Frame: as for outcome 1
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number; unit: Subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Subjects
  Any AE | 13 | 5
  Any SAE | 1 | 0

4. Secondary Outcome: Incidence Rates of Musculoskeletal Adverse Events by Primary System Organ Class (SOC) and Preferred Term
Description: Musculoskeletal adverse events were classified as following SOCs (preferred terms): "injury, poisoning and procedural complications" (forearm fracture, joint injury, ligament sprain, muscle strain) "musculoskeletal and connective tissue disorders" (arthralgia, joint swelling, musculoskeletal pain, myalgia). Incidence rates were reported as percentage of subjects categorized under preferred terms.
Time Frame: as for outcome 1
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Percentage of subjects
  Forearm fracture | 0.3 [0.01 to 1.84] | 0 [0 to 2.43]
  Joint injury | 0 [0 to 1.22] | 0.7 [0.02 to 3.66]
  Ligament sprain | 0.3 [0.01 to 1.84] | 0.7 [0.02 to 3.66]
  Muscle strain | 0 [0 to 1.22] | 0.7 [0.02 to 3.66]
  Arthralgia | 3 [1.38 to 5.6] | 1.3 [0.16 to 4.73]
  Joint swelling | 0 [0 to 1.22] | 0.7 [0.02 to 3.66]
  Musculoskeletal pain | 1 [0.21 to 2.88] | 0 [0 to 2.43]
  Myalgia | 0.3 [0.01 to 1.84] | 0 [0 to 2.43]

5. Secondary Outcome: Heart Rate Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Beats per minute (bpm)
  Day 1: Pre-dose (N= 300, 150) | 93.4 (19.1) | 90.4 (16.9)
  Change at Day 1 ((N= 294, 148) | 2.8 (9.7) | 0.3 (6.9)
  Day 3: Pre-dose (N= 293, 146) | 84.3 (17.2) | 82.6 (16.2)
  Change at Day 3 (N= 290, 146) | 1 (8.9) | -0.9 (7.1)

6. Secondary Outcome: PR Interval Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: The PR interval is defined as the period that extends from the onset of atrial depolarization (beginning of the P wave) until the onset of ventricular depolarization. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 299, 150) | 136.8294 (18.3554) | 140.5933 (20.5113)
  Change at Day 1 ( N= 292, 148) | 0.7123 (8.2587) | -0.0203 (8.5631)
  Day 3: Pre-dose (N= 293, 146) | 139.4915 (17.3258) | 139.5685 (20.8174)
  Change at Day 3 (N= 289, 146) | 1.5813 (9.2143) | 1.5616 (9.9322)

7. Secondary Outcome: RR Interval Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: The RR interval refers to the respective time interval in the Electrocardiogram. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 300, 150) | 670.7567 (142.6153) | 689.3067 (145.5957)
  Change at Day 1 (N= 294, 148) | -20.6429 (74.3401) | -3.4797 (56.9955)
  Day 3: Pre-dose (N= 293, 146) | 740.4778 (149.0964) | 754.6027 (150.1203)
  Change at Day 3 (N= 290, 146) | -9.2862 (77.7582) | 10.5137 (67.1124)

8. Secondary Outcome: QRS Interval Changes in Electrocardiogram (ECG) Profiles From Predose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: The QRS interval represents the time it takes for ventricular depolarization to occur. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 300, 150) | 89.0333 (7.8279) | 88.8067 (7.9264)
  Change at Day 1 (N= 294, 148) | 0.119 (4.3799) | 1.223 (4.2568)
  Day 3: Pre-dose (N= 293, 146) | 89.2423 (8.0196) | 89.3904 (7.8198)
  Change at Day 3 (N= 289, 146) | 0.2768 (4.123) | 0.2877 (3.1687)

9. Secondary Outcome: QT Interval Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: The QT interval is the period that extends from the beginning of ventricular depolarization until the end of ventricular repolarization. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 298, 150) | 341.1812 (33.9858) | 344.2333 (33.5494)
  Change at Day 1 (N= 290, 148) | 2.5828 (15.213) | 1.1149 (11.5744)
  Day 3: Pre-dose (N= 292, 146) | 358.3082 (34.0504) | 356.5822 (35.6653)
  Change at Day 3 (N= 287, 146) | 6.0906 (16.1875) | 3.1644 (11.9586)

10. Secondary Outcome: Corrected QT (QTc) Interval Calculated (Calc) Bazett Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: QTc interval Calc Bazett represent the interval corrected for heart rate (QTc) milliseconds (msec) which was calculated by Bazett's method. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 298, 150) | 419.5872 (19.3278) | 417.34 (18.5718)
  Change at Day 1 (N= 290, 148) | 9.731 (14.2961) | 2.2905 (14.2544)
  Day 3: Pre-dose (N= 292, 146) | 419.2055 (16.6815) | 412.7945 (17.0075)
  Change at Day 3 (N= 287, 146) | 9.2509 (16.8132) | 1 (12.5346)

11. Secondary Outcome: Corrected QT (QTc) Interval Calculated (Calc) Fridericia Changes in Electrocardiogram (ECG) Profiles From Pre-dose to Post-dose on Treatment Day 1 and Treatment Day 3
Description: QTc interval Calc Fridericia represent the interval corrected for heart rate (QTc) msec which was calculated by Fridericia's method. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
milliseconds
  Day 1: Pre-dose (N= 298, 150) | 391.1846 (19.1574) | 390.9467 (18.4339)
  Change at Day 1 (N= 290, 148) | 7.0724 (11.3219) | 1.9122 (11.3058)
  Day 3: Pre-dose (N= 292, 146) | 397.3767 (17.2179) | 392.6918 (18.8144)
  Change at Day 3 (N= 287, 146) | 8.115 (13.5805) | 1.774 (9.3328)

12. Secondary Outcome: Potentially Clinically Significant Electrocardiogram (ECG) QTc Interval Prolongation - by QTc Interval Calc Fridericia Correction on Treatment Day 1 and During Therapy Day 3
Description: A significant QTc prolongation was considered when the QTc value was more than (>) upper limit of normal (ULN) range or was prolonged for 30 msec or 60msec in comparison with the pre-treatment value measured on Day 1. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively. Percentage of subjects with potentially clinically significant ECG data was reported.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Percentage of subjects
  Day1: Pre-dose QTcCalcFridericia>ULN (N= 300, 150) | 0.7 (19.1574) | 1.3 (18.4339)
  Day1: Post-dose QTcCalcFridericia>ULN (N= 297,148) | 3 (11.3219) | 2 (11.3058)
  Day1: Post-dose >30 ms from pre-dose (N= 297,148) | 2 (17.2179) | 0 (18.8144)
  Day1: Post-dose >60 ms from pre-dose (N= 297,148) | 0.3 (13.5805) | 0 (9.3328)
  Day3: Pre-dose QTcCalcFridericia>ULN (N= 293, 146) | 1.4 | 1.4
  Day3: Post-dose QTcCalcFridericia>ULN (N= 291,148) | 9.6 | 1.4
  Day3: Post-dose >30 ms from pre-dose (N= 291,148) | 17.9 | 3.4
  Day3: Post-dose >60 ms from pre-dose (N= 291,148) | 1.7 | 0.7

13. Secondary Outcome: Potentially Clinically Significant Electrocardiogram (ECG) QTc Interval Prolongation - by QTc Calc Bazett Correction on Treatment Day 1 and During Therapy Day 3
Description: A significant QTc prolongation was considered when the QTc value was more than ULN range or was prolonged for 30 msec or 60msec in comparison with the pre-treatment value measured on Day 1. "N" signifies subjects who were evaluable for the specified parameter for each arm, respectively. Percentage of subjects with potentially clinically significant ECG data was reported.
Time Frame: Baseline (Pre-dose), Day 1, Day 3
Population: Safety analysis set; All subjects (N= 451) treated with at least one dose of study medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 301 | 150
Percentage of subjects
  Day1: Pre-dose QTc Calc Bazett > ULN (N= 300, 150) | 7.7 | 2.7
  Day1: Post-dose QTc Calc Bazett > ULN (N= 297,148) | 16.2 | 4.1
  Day1: Post-dose >30 ms from pre-dose (N= 297,148) | 5.4 | 0
  Day1: Post-dose >60 ms from pre-dose (N= 297,148) | 0 | 0
  Day3: Pre-dose QTc Calc Bazett > ULN (N= 293, 146) | 3.8 | 1.4
  Day3: Post-dose QTc Calc Bazett > ULN (N= 291,148) | 15.5 | 3.4
  Day3: Post-dose >30 ms from pre-dose (N= 291,148) | 9.6 | 2
  Day3: Post-dose >60 ms from pre-dose (N= 291,148) | 0.7 | 0.7

14. Secondary Outcome: Clinical Response at Test-of-Cure (TOC) Visit
Description: Clinical responses were graded as clinical cure, failure or indeterminate. 'Clinical cure' defined as a resolution or sufficient improvement of clinical signs and symptoms related to the infection; 'failure' defined as a reappearance of the signs and symptoms of the original infection, or wound infection requiring further systemic antimicrobial therapy; 'indeterminate' defined as those subjects in whom a clinical assessment was not possible to determine (due to early withdrawal from the study because of adverse events, protocol violation, withdrawn consent). Percentage of subjects with clinical response at TOC were reported.
Time Frame: 28 to 42 days
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 297 | 150
Percentage of subjects
  Clinical Cure | 86.2 | 95.3
  Clinical Failure | 5.7 | 2
  Indeterminate | 8.1 | 2.7

15. Secondary Outcome: Bacteriological Response at Test-of-Cure (TOC) Visit
Description: Bacteriological responses were graded as presumed persistence, presumed eradication or indeterminate.
  'Presumed persistence' was applicable for subjects judged to be clinical failures, and appropriate culture material is not available for evaluation; 'presumed eradication' defined as the absence of appropriate culture material for evaluation because the subject has clinically responded and invasive procedures are not warranted; índeterminate' was applicable when the bacteriological response to the study drug was not valid for any reason (eg, pre-treatment culture was negative or culture was not obtained when material was available and the subject was not judged a clinical failure). Percentage of subjects with bacteriological response at TOC were reported.
Time Frame: 28 to 42 days
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 249 | 136
Percentage of subjects
  Presumed Persistence | 6.8 | 2.2
  Presumed Eradication | 84.7 | 94.9
  Indeterminate | 8.4 | 2.9

16. Secondary Outcome: Clinical Response at Test-of-Cure (TOC) Visit in Subjects With Bacteriologically Confirmed Complicated Intra-abdominal Infection (cIAI)
Description: as for outcome 14
Time Frame: 28 to 42 days
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 297 | 150
Percentage of subjects
  Clinical Cure | 86.2 | 95.3
  Clinical Failure | 5.7 | 2
  Indeterminate | 8.1 | 2.7

17. Secondary Outcome: Clinical Response at a 'During Therapy' Visit
Description: Clinical responses during therapy visit were graded as clinical improvement, clinical failure, or indeterminate. Clinical improvement defined as a reduction in the severity and/or the number of signs and symptoms of infection; 'clinical failure' defined as a failure to respond or insufficient lessening of the signs and symptoms of infection requiring a modification or addition of antibacterial therapy.
  'Indeterminate' defined as those subjects in whom a clinical assessment is not possible to determine (eg, due to early withdrawal from the study because of adverse events, protocol violation, withdrawn consent, receipt of an effective concomitant antibacterial for an indication other than the study indication and receipt of less than 3 full days of study drug, etc). Percentage of subjects with clinical response during therapy visit were reported.
Time Frame: Day 3 to Day 5
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 299 | 148
Percentage of subjects
  Clinical Improvement | 94.3 | 98
  Clinical Failure | 1 | 0.7
  Indeterminate | 4.7 | 1.4

18. Secondary Outcome: Bacteriological Response at a 'During Therapy' Visit
Description: Bacteriological response during therapy were graded as presumed persistence, presumed eradication, or indeterminate'Presumed persistence' is applicable for subjects judged to be clinical failures and appropriate culture material is not available for evaluation;'presumed eradication' is defined as the absence of appropriate culture material for evaluation because the subject has clinically responded (with a response as a resolution or cure) and invasive procedures are not warranted; 'indeterminate is applicable when the bacteriological response to the study drug is not valid for any reason (eg, pretreatment culture was negative or culture was not obtained when material was available and the subject is not judged a clinical failure). Percentage of subjects with bacteriological response during therapy visit were reported
Time Frame: Day 3 to Day 5
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 249 | 134
Percentage of subjects
  Presumed Persistence | 1.2 | 0.7
  Presumed Eradication | 95.6 | 97.8
  Indeterminate | 3.2 | 1.5

19. Secondary Outcome: Clinical Response at the End-of-Treatment (EOT) Visit
Description: Clinical responses at EOT were graded as resolution, failure, or indeterminate. 'Resolution' defined as a disappearance of signs and symptoms related to the infection or sufficient improvement of clinical signs and symptoms related to the infection and the subject does not require any further antibiotic therapy or surgical intervention; 'failure' defined as worsening or insufficient lessening of the signs and symptoms of infection requiring a modification or addition of antibacterial therapy; 'indeterminate' is defined as those subjects in whom a clinical assessment is not possible to determine (eg, due to early withdrawal from the study because of adverse events, protocol violation, withdrawn consent; receipt of less than 3 full days of study drug; receipt of an effective concomitant antibacterial for an indication other than study indication; etc). Percentage of subjects with clinical response at EOT were reported.
Time Frame: Day 5 to Day 14
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 283 | 148
Percentage of subjects
  Resolution | 92.2 | 98
  Clinical Failure | 4.6 | 0.7
  Indeterminate | 3.2 | 1.4

20. Secondary Outcome: Bacteriological Response at the End of Treatment (EOT) Visit
Description: Bacteriological response at EOT were grades as presumed persistence, presumed eradication or indeterminate. 'presumed persistence' was applicable for subjects judged to be clinical failures and appropriate culture material is not available for evaluation; 'presumed eradication' defined as the absence of appropriate culture material for evaluation because the subject has clinically responded (with a response as a resolution or cure) and invasive procedures are not warranted; 'indeterminate' is applicable when the bacteriological response to the study drug was not valid for any reason (eg, pretreatment culture was negative or culture was not obtained when material was available and the subject was not judged a clinical failure). Percentage of subjects with bacteriological response at EOT were reported.
Time Frame: Day 5 to Day 14
Population: Safety analysis set with subjects evaluable for this outcome
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Number analyzed (Participants) | 237 | 134
Percentage of subjects
  Presumed Persistence | 5.5 | 0.7
  Presumed Eradication | 91.1 | 97.8
  Indeterminate | 3.4 | 1.5

ADVERSE EVENTS:
Time Frame: All AEs and SAE were recorded from treatment start to test of cure visit; musculoskeletal AEs were recorded up to 1 year post-end of treatment (EOT) visit; subjects with musculoskeletal AEs 1 year after EOT were followed up to 5 years or until resolution.
Groups:
- Moxifloxacin (Avelox, BAY12-8039): Subjects randomized to the moxifloxacin arm of this study received intravenous moxifloxacin plus ertapenem placebo (0.9 % NaCl solution) for a minimum of 3 days and, if switched to oral treatment, PO moxifloxacin plus PO amoxicillin/clavulanate placebo. Total treatment duration is 5-14 days.
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Comparator Ertapenem
Serious Adverse Events (participants affected / at risk) | 20/301 | 6/150
Other Adverse Events (participants affected / at risk) | 127/301 | 63/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (Avelox, BAY12-8039) (N=301) | Comparator Ertapenem (N=150)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 3 (3) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecalith (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (3) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (Avelox, BAY12-8039) (N=301) | Comparator Ertapenem (N=150)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 20 (22) | 12 (12)
Pyrexia (General disorders) | 6 (6) | 4 (4)
Infusion site phlebitis (General disorders) | 4 (6) | 0 (0)
Wound infection (Infections and infestations) | 13 (13) | 6 (6)
Wound complication (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 26 (26) | 14 (14)
Postoperative wound complication (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 16 (16) | 10 (10)
Incision site inflammation (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 28 (31) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 2 (2)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (36) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Abdominal cavity drainage (Surgical and medical procedures) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12/18 months after database lock at the earliest.

* Bayer will have up to 30/45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).
* No publication of single center data should be done prior of publication if multi-center data.